CLINICAL TRIAL: NCT06272162
Title: Locally Advanced Pancreatic Cancer After Systemic Therapy: Ablative MR-guided Radiotherapy, a Randomized Controlled Trial
Brief Title: Locally Advanced Pancreatic Cancer After Systemic Therapy: Ablative MR-guided Radiotherapy
Acronym: LAPSTAR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Amsterdam UMC, location VUmc (Other); Radboud University Medical Center (Other); Catharina Ziekenhuis Eindhoven (Other); Centre for Human Drug Research, Netherlands (Other); Dutch Pancreatic Cancer Group (DPCG) (Unknown)
Responsible Party: Principal Investigator, Lois Daamen, Prinipal Investigator, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL85622.041.24; 15030 (Other Grant/Funding Number: KWF); 23U-0725 (Other: NedMec)
Record Dates: First submitted 2024-01-08; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Locally Advanced Pancreatic Adenocarcinoma
Keywords: MR guided radiation therapy

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Patients in the intervention arm will receive locally ablative stereotactic MRgRT in addition to standard of care, consisting of 5 times 10 Gy MR guided radiotherapy.
  Interventions: Radiation: MR guided radiotherapy
- Control arm (No Intervention): Patients randomized to the control arm will continue standard of care as described without additional local treatment.

INTERVENTIONS:
Radiation: MR guided radiotherapy — 5 fractions of 10 Gray MRgRT in addition to standard of care
  Arms: Intervention arm

SUMMARY:
A randomized controlled trial comparing the effect of local ablative MR-guided radiotherapy (MRgRT) after systemic therapy with current standard treatment alone, on health-related quality of life in patients with locally advanced pancreatic cancer (LAPC).

DETAILED DESCRIPTION:
Rationale: About 40% of patients with pancreatic cancer are diagnosed with locally advanced pancreatic cancer (LAPC). Recommended treatment consists of chemotherapy to prevent disease dissemination and prolong survival. Nevertheless, local tumor growth often causes severe morbidity, including pain, gastrointestinal obstruction, and malnutrition. This has a substantial negative impact on health-related quality of life (HRQoL). Eventually, one-third of patients die due to local tumor growth rather than from systemic disease spread. For palliation of symptoms and improved local tumor control, potentially prolonging survival, minimally-invasive ablative therapies may be effective. Online adaptive stereotactic Magnetic Resonance-guided radiotherapy (MRgRT) is an innovative treatment modality that enables high-precision ablative radiotherapy for pancreatic tumors. This potentially improves RT efficacy without increasing the risk of RT-related toxicity. Consequently, MRgRT holds promise for the treatment of pancreatic cancer.

Objective: To investigate the efficacy of stereotactic MRgRT on HRQoL deterioration-free survival, including death as an event, in patients with LAPC after systemic chemotherapy.

Study design: Nationwide randomized controlled trial (1:1 randomization).

Study population: Patients with LAPC according to Dutch Pancreatic Cancer Group (DPCG) criteria who are not eligible for tumor resection after at least two months of chemotherapy (sample size 150 patients). Also, patients with LAPC who are eligible but choose to refrain from chemotherapy and/or surgery can participate in this trial.

Intervention: Patients in the intervention arm receive 50Gy MRgRT in five fractions over two weeks in one of the four Consortium Centers, followed by standard care, either consisting of continuation of chemotherapy or best supportive care. Patients in the control arm continue standard care without ablative MRgRT.

Main study endpoints: The primary outcome is HRQoL deterioration-free survival from the time of randomization, defined as the Time Until Definitive Deterioration (TUDD) including death as an event. HRQoL is evaluated using the EORTC QLQ-C30 Summary Score. The TUDD is defined as a 10-point minimal clinically important difference compared to baseline, with no further improvement of ≥10 points afterwards. All patients will be offered home monitoring using the Trial@home platform to decrease the burden of trial participation.

ELIGIBILITY:
Inclusion Criteria:

* Pathology proven pancreatic ductal adenocarcinoma (PDAC);
* At least two (preferably four) months systemic therapy with (m)FOLFIRINOX and/or gemcitabine + nab-paclitaxel; or eligibility for chemotherapy but no initiation of chemotherapy based on patients' wish;
* No option for surgical resection, either because anatomical irresectability based on the surgeon's judgement (assessed on imaging or during explorative laparotomy) and/or frailty (unfit for surgery or chemotherapy) and/or no surgery based on patient's wish.
* No evidence of distant metastatic disease progression, evaluated by CT Thorax / Abdomen / Pelvis and/or PET-CT scan;
* Performance status WHO 0-2.

Exclusion Criteria:

* Contra-indications for MRI or CT with an intravenous contrast agent according to the protocol of the local radiology and/or radiotherapy departments

  * Contraindications for MRgRT, as determined by the involved expert radiation oncologists of the Consortium
  * <18 years old
  * Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
HRQoL deterioration-free survival | Through study completion, an average of 18 months
  HRQoL deterioration-free survival is defined as the Time Until Definitive Deterioration (TUDD) including death from any cause, calculated from the time of randomization. HRQoL is primarily assessed using the EORTC QLQ-C30 (version 3.0) Summary Score.

SECONDARY OUTCOMES:
Overall survival | From the date of LAPC diagnosis untill either death from any cause or last follow-up, whichever came first, assessed up to 18 months
  The time interval between LAPC diagnosis and either death from any cause or last follow-up
Patient reported Quality of Life EORTC QLQ-PAN26 | At baseline and at 2,4, weeks and subsequently every 2 months. Assessed through study completion, up to 18 months
  Part of the Patient Reported Outcome Measures (PROMs) using EORTC QLQ-PAN26
Patient reported Quality of Life EORTC QLQ-C30 | At baseline and at 2,4, weeks and subsequently every 2 months. Assessed through study completion, up to 18 months
  Part of the Patient Reported Outcome Measures (PROMs) using EORTC QLQ-C30
Patient reported Quality of Life EQ5D-5L | At baseline and at 2,4, weeks and subsequently every 2 months. Assessed through study completion, up to 18 months
  Part of the Patient Reported Outcome Measures (PROMs) using EQ5D-5L
The need of subsequent treatments | Through study completion, an average of 18 months
  To assess continuation of systemic therapy and/or administration of subsequent treatments (e.g., surgery, second-line systemic treatment, experimental treatment in clinical studies etc.), recommendations from multidisciplinary team meetings, reasons for refraining from recommended therapy, and reasons for discontinuation of therapy (i.e., start of best supportive care)
Treatment response assessed on CT-imaging (graded according to RECIST guidelines) | with available imaging during 18 months follow-up
  To assess tumor response on imaging according to RECIST criteria in patients who received imaging procedures during follow-up (no part of the trial follow-up)
CA 19.9 response | Through study completion, an average of 18 months
  To assess serum CA 19-9 response in patients in whom serum CA 19-9 is measured (no part of the trial follow-up)
Trial@home monitoring related outcome: feasibility Withings Steel HR smartwatch | Through study completion, an average of 18 months
  To assess the feasibility of the Trial@home monitoring via the Withings Steel HR smartwatch for home monitoring of pancreatic cancer patients.
  Compliance Withings Steel HR smartwatch (wear-time): amount of time (hours) in a day that the participant wears the smartwatch. This is calculated by the amount of time the device registers a heart rate. Patients wearing the device for >50% of the observation period will be considered as feasible.
Trial@home monitoring related outcome: feasibility Body+ scale | Through study completion, an average of 18 months
  To assess the feasibility of the Trial@home monitoring via the Body+ scale for home monitoring of pancreatic cancer patients.
  Compliance rates Body+ scale: compliance with weekly weight measurements is calculated by the number of completed weight measurements divided by the total amount of weeks in the observation period. A compliance rate of at least 75% will be considered as feasible.
Trial@home monitoring related outcome: feasibility Whitings Sleep | Through study completion, an average of 18 months
  To assess the feasibility of the Trial@home monitoring via the Whitings Sleep for home monitoring of pancreatic cancer patients.
  Compliance Whitings Sleep: compliance with daily sleep monitoring is calculated by the number of nights sleep is measured. A compliance rate of at least 75% nights per week will be considered as feasible.
Trial@home monitoring related outcome: feasibility ePRO application | Through study completion, an average of 18 months
  To assess the feasibility of the Trial@home monitoring via the ePRO application for home monitoring of pancreatic cancer patients.
  Compliance questionnaires through the ePROapplication: A compliance rate of at least 75% from the scheduled assessments will be considered as feasible.
Trial@home monitoring related outcome: digital biomarkers | Through study completion, an average of 18 months
  To exploratively generate digital biomarkers and quantify the correlation between data obtained from the Trial@home platform (Withings Steel HR smartwatch, a Withings Body+ Scale, a Withings Sleep, ePRO) and clinical endpoints (e.g., unplanned hospitalizations, early signs of adverse events, clinical deterioration, performance status, quality of life)
Intervention arm related outcome toxicity | Through study completion, an average of 18 months
  To assess acute (3 months) RT-related toxicity measured from the start of MRgRT, according to CTCAE v527
Intervention arm related outcome, completion of therapy | Through study completion, an average of 18 months
  To assess completion of therapy
Intervention arm related outcome diffusion weighted images | Through study completion, an average of 18 months
  To assess correlation of diffusion weighted images at each treatment fraction and the possible correlation with outcomes for patients treated on a 1.5T MR-Linac

CONTACTS AND LOCATIONS:
Overall Officials: L. A. Daamen, MD, PhD, Principal Investigator — Regional Academic Cancer Center Utrecht (RACU); M P.W. Intven, MD, PhD, Principal Investigator — Regional Academic Cancer Center Utrecht (RACU); A. M.E. Bruynzeel, MD, PhD, Principal Investigator — Amsterdam University Medical Center, VUmc; H. D. Heerkens, MD, PhD, Principal Investigator — Radboud University Medical Center; H. M.U. Peulen, MD, PhD, Principal Investigator — Catharina Ziekenhuis Eindhoven; J. J. Bosch, Principal Investigator — Centre of Human Drug Research
Locations (4):
- Netherlands (4):
  - Catharina Hospital, Eindhoven, North Brabant
  - Amsterdam University Medical Center, VUmc, Amsterdam, North Holland
  - Radboud University Medical Center, Nijmegen
  - University Medical Center Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
De-dentified data generated during the LAPSTAR trial will be made available to other researchers upon request from L.A. Daamen
Supporting Information: Study Protocol
Access Criteria: upon request